CLINICAL TRIAL: NCT01885624
Title: Open Label Phase 1 Pharmacokinetics and Tolerability Study of Single TAB08 Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theramab LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAB08/HS/R1
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Adult Healthy Volunteers
Keywords: TAB08; healthy volunteers
MeSH Terms: interventions — TGN-1412

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAB08 (Experimental): Single TAB08 i.v. infusion
  Interventions: Biological: TAB08

INTERVENTIONS:
Biological: TAB08 — monoclonal antibody

SUMMARY:
The purpose of this study is to assess safety and tolerability of ascending dosed of TAB08 after single i.v. infusion to the adult healthy volunteers. Additionally were assessed infusion speed tolerability, pharmacokinetics and pharmacodynamics of TAB08 after single i.v. infusion and to explore TAB mechanism-of-action biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult man aged from 18 to 40 years, who agreed to use adequate contraception.
* Body mass is at least 60 kg and BMI is within 20-27
* Volunteer is in good physical and mental health, as per his medical history and assessment results
* Volunteer's laboratory values are normal (or not clinically significant as per Investigator discretion) at screening, including baseline cytokines levels as per RESTORE test results
* Volunteer has signed the informed concent.

Exclusion Criteria:

* Any chronic or relapsing illness in the medical history
* Any abnormal assessment or laboratory result at screening, which is clinically significant as per Investigator discretion
* Active tuberculosis at the time of screening
* Any acute illness at the time of study enrollment
* Any blood donation within 4 weeks before Study Day 1
* Positive result for HBsAG, Hepatitis C, HIV
* Continuous use af any medications
* Use of any medications within 72 hours before study drug infusion
* Use of an investigational treatment within 4 weeks before screening, or within a period of 5 half-lives of the investigational treatment, whichever is longer
* High inflammatory cytokines levels as per RESTORE test results after ex vivo PBMC testing

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity in every dose cohort | From study drug infusion (Day 1) untill the end of study (Day 71/141)

CONTACTS AND LOCATIONS:
Overall Officials: Olga B Ershova, Prof., Principal Investigator — Clinical Emergency Hospital of Yaroslavl
Locations (1):
- Clinical Emergency Hospital of Yaroslavl, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No